CLINICAL TRIAL: NCT02243046
Title: The Clinical Investigation of a Zinc Based Toothpaste as Compared to a Triclosan Based Toothpaste and Colgate Fluoride Toothpaste in Reducing Established Plaque and Gingivitis - a Six-month Study.
Brief Title: The Clinical Investigation of a Zinc Based Toothpaste in Reducing Plaque and Gingivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-2014-11-PG-ZNPTCN-ED
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2015-07

CONDITIONS: Dental Plaque and Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis | interventions — hydrated silica gel-based toothpaste

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control toothpaste (Placebo Comparator): 1450 ppm Fluoride toothpaste
  Interventions: Drug: Control toothpaste
- Experimental toothpaste (Experimental): 1450 ppm sodium fluoride toothpaste with a zinc base
  Interventions: Drug: Experimental toothpaste
- Active comparator (Active Comparator): 1450 ppm sodium fluoride/triclosan toothpaste
  Interventions: Drug: Active Comparator

INTERVENTIONS:
Drug: Control toothpaste — 1450 ppm fluoride toothpaste control - Subjects will brush their whole mouth with the control toothpaste 2 times/day for 1 minute each time and rinse with water after brushing. This daily brushing routine will continue for the six (6) month study.
  Other Names: Max Fresh toothpaste
  Arms: Control toothpaste
Drug: Experimental toothpaste — 1450 ppm sodium fluoride/zinc base toothpaste - Subjects will brush their whole mouth with a fluoride/zinc toothpaste 2 times/day for 1 minute each time and rinse with water after brushing. This daily brushing routine will continue for the six (6) month study.
  Arms: Experimental toothpaste
Drug: Active Comparator — 1450 ppm sodium fluoride/triclosan toothpaste - Subjects will brush their whole mouth with this toothpaste 2 times/day for 1 minute each time and rinse with water after brushing. This daily brushing routine will continue for the six (6) month study.
  Other Names: Total toothpaste
  Arms: Active comparator

SUMMARY:
This is a six (6) month, double-blind, parallel, controlled clinical trial utilizing one hundred and sixty (160) adults to evaluate the reduction of dental plaque and gingivitis.

ELIGIBILITY:
Inclusion Criteria

1. Subjects, ages 18-70, inclusive.
2. Availability for the six-month duration of the clinical research study.
3. Good General health.
4. Minimum of 20 uncrowned permanent natural teeth (excluding third molars).
5. Initial gingivitis index of at least 1.0 as determined by the use of the Loe and Silness Gingival Index.
6. Initial plaque index of at least 1.5 as determined by the use of the Quigley and Hein Plaque Index (Turesky Modification).
7. Signed Informed Consent Form.

Exclusion Criteria

1. Presence of orthodontic bands.
2. Presence of partial removable dentures.
3. Tumor(s) of the soft or hard tissues of the oral cavity.
4. Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone).
5. Five or more carious lesions requiring immediate restorative treatment.
6. Antibiotic use any time during the one-month period prior to entry into the study.
7. Participation in any other clinical study or test panel within the one month prior to entry into the study.
8. Dental prophylaxis during the past two weeks prior to baseline examinations.
9. History of allergies to oral care/personal care consumer products or their ingredients.
10. On any prescription medicines that might interfere with the study outcome.
11. An existing medical condition that prohibits eating or drinking for periods up to 4 hours.
12. History of alcohol or drug abuse.
13. Pregnant or lactating subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Spa Dental, Santo Domingo, Dominican Republic

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Toothpaste | Experimental Toothpaste | Active Comparator
Started | 55 | 54 | 53
3 Month | 54 (1 subject didn't return for 3 month clinic visit) | 53 (1 subject didn't return for 3 month clinic visit) | 51 (2 subjects didn't return for 3 month clinic visit)
6 Month | 54 | 53 | 49 (2 subjects didn't return for 6 month clinic visit)
Completed | 54 | 53 | 49
Not Completed | 1 | 1 | 4
Not completed — Lost to Follow-up | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Toothpaste | Experimental Toothpaste | Active Comparator | Total
Number analyzed (Participants) | 55 | 54 | 53 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.52 (10.99) | 30.92 (9.82) | 30.39 (13.47) | 30.62 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 31 | 28 | 93
  Male | 21 | 23 | 25 | 69
Region of Enrollment [Number; unit: participants]
  Dominican Republic | 55 | 54 | 53 | 162

OUTCOME MEASURES:

1. Primary Outcome: Gingivitis Scores
Description: Gingivitis scale (Loe & Silness Gingival Index) Units on a scale 0 to 3 (0 = no inflammation, 1 = Mild inflammation-slight change in color and little change in texture 2 = Moderate inflammation-moderate glazing, redness, edema and hypertrophy. Tendency to bleed upon probing. 3 = Severe inflammation-marked redness and hypertrophy. Tendency to spontaneous bleeding)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Toothpaste | Experimental Toothpaste | Active Comparator
Number analyzed (Participants) | 55 | 54 | 53
units on a scale | 1.48 (0.23) | 1.57 (0.28) | 1.49 (0.20)
Statistical Analysis 1: Comparison: Control Toothpaste vs Experimental Toothpaste vs Active Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.091, ANOVA

2. Primary Outcome: Gingivitis Scores
Description: as for outcome 1
Time Frame: 3 months (from Baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Toothpaste | Experimental Toothpaste | Active Comparator
Number analyzed (Participants) | 54 | 53 | 51
units on a scale | 1.46 (0.19) | 1.33 (0.23) | 1.25 (0.18)
Statistical Analysis 1: Comparison: Control Toothpaste vs Experimental Toothpaste vs Active Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.001, ANCOVA

3. Primary Outcome: Gingivitis Scores
Description: as for outcome 1
Time Frame: 6 months (from Baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Toothpaste | Experimental Toothpaste | Active Comparator
Number analyzed (Participants) | 54 | 53 | 49
units on a scale | 1.44 (0.20) | 1.23 (0.23) | 1.19 (0.17)
Statistical Analysis 1: Comparison: Control Toothpaste vs Experimental Toothpaste vs Active Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.001, ANCOVA

4. Primary Outcome: Dental Plaque Scores
Description: Dental Plaque (Quigley-Hein, Turesky Modification Index) Units on a scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque, 3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Toothpaste | Experimental Toothpaste | Active Comparator
Number analyzed (Participants) | 55 | 54 | 53
units on a scale | 2.91 (0.24) | 2.95 (0.29) | 2.90 (0.20)
Statistical Analysis 1: Comparison: Control Toothpaste vs Experimental Toothpaste vs Active Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p = 0.571, ANOVA

5. Primary Outcome: Dental Plaque Scores
Description: as for outcome 4
Time Frame: 3 months (from Baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Toothpaste | Experimental Toothpaste | Active Comparator
Number analyzed (Participants) | 54 | 53 | 51
units on a scale | 2.59 (0.29) | 2.16 (0.53) | 2.10 (0.36)
Statistical Analysis 1: Comparison: Control Toothpaste vs Experimental Toothpaste vs Active Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.001, ANCOVA

6. Primary Outcome: Dental Plaque Scores
Description: as for outcome 4
Time Frame: 6 months (from Baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Toothpaste | Experimental Toothpaste | Active Comparator
Number analyzed (Participants) | 54 | 53 | 49
units on a scale | 2.47 (0.42) | 1.82 (0.45) | 1.75 (0.39)
Statistical Analysis 1: Comparison: Control Toothpaste vs Experimental Toothpaste vs Active Comparator; The null hypothesis states that there is no difference between groups; Test type: Superiority or Other; p < 0.001, ANCOVA

ADVERSE EVENTS:
Time Frame: Baseline, 3 and 6 months
Groups:
- Active Comparator: 1450 ppm sodium fluoride/triclosan toothpaste Active Comparator: 1450 ppm sodium fluoride/triclosan toothpaste - Subjects will brush their whole mouth with this toothpaste 2 times/day for 1 minute each time and rinse with water after brushing. This daily brushing routine will continue for the six (6) month study.
Arm/Group | Control Toothpaste | Experimental Toothpaste | Active Comparator
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/54 | 0/53
Other Adverse Events (participants affected / at risk) | 0/55 | 0/54 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days